CLINICAL TRIAL: NCT04522050
Title: A Multicenter and Prospective Clinical Trial of Gemcitabine-based Induction Chemotherapy Combined With Concurrent Chemoradiotherapy in Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Gemcitabine-based Induction Chemotherapy Combined With Concurrent Chemoradiotherapy in Locally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qi Zeng, Principal Investigator, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.TJZLK.111
Record Dates: First submitted 2020-08-15; First posted 2020-08-21 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-06

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Chemoradiotherapy; Gemcitabine

STUDY DESIGN:
Intervention Model Description: The initial dose of gemcitabine is 25mg/m² once a week for 6 times. The patients are divided into 9 groups (25mg/m², 50mg/m², 100mg/m², 200mg/m², 300mg/m², 350mg/m², 400mg/m², 450mg/m², 500mg/m²) with 6 patients in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction chemotherapy + IMRT and concurrent gemcitabine (Other): Patients receive gemcitabine (1000mg/m² d1,8) and cisplatin (80mg/m²,d1) every 3weeks for 2 cycles before radiotherapy, and then receive intensity modulated radiotherapy (IMRT) concurrently with gemcitabine. The initial dose of gemcitabine is 25mg/m² once a week for 6 times. Patients are divided into 9 groups (25mg/m², 50mg/m², 100mg/m², 200mg/m², 300mg/m², 350mg/m², 400mg/m², 450mg/m², 500mg/m²) with 6 patients in each group.
  Interventions: Drug: Gemcitabine combined with cisplatin induction chemotherapy; Drug: concurrent chemoradiotherapy with gemcitabine

INTERVENTIONS:
Drug: Gemcitabine combined with cisplatin induction chemotherapy — Patients receive gemcitabine (1000mg/m² d1,8) and cisplatin (80mg/m², d1) every 3 weeks for 2 cycles before radiotherapy. And then intensity modulated radiotherapy (IMRT) is given a total dose of GTVnx 70Gy, GTVnd 66Gy, CTV1 60Gy and CTV2 54Gy for 33 times in total, concurrently with gemcitabine. The initial dose of gemcitabine is 25mg/m² once a week for 6 times. The patients are divided into 9 groups (25mg/m², 50mg/m², 100mg/m², 200mg/m², 300mg/m², 350mg/m², 400mg/m², 450mg/m², 500mg/m²) with 6 patients in each group.
  Other Names: concurrent chemoradiotherapy with gemcitabine
Drug: concurrent chemoradiotherapy with gemcitabine — followed by concurrent gemcitabine chemoradiotherapy

SUMMARY:
Researchers conduct the clinical trial (gemcitabine combined with cisplatin induction chemotherapy followed by concurrent chemoradiotherapy with gemcitabine for locally advanced nasopharyngeal carcinoma) to evaluate the safety and effectiveness of gemcitabine in patients with locally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Diagnosed as locally advanced nasopharyngeal carcinoma (stage III-IV), and pathologically confirmed as a differentiated or undifferentiated non-keratinizing nasopharyngeal carcinoma, the patient is eligible to participate in the study. Patients receive gemcitabine (1000mg/m² d1,8) and cisplatin (80mg/m², d1) every 3 weeks for 2 cycles before radiotherapy. And then intensity modulated radiotherapy (IMRT) is given a total dose of GTVnx 70Gy, GTVnd 66Gy, CTV1 60Gy and CTV2 54Gy for 33 times in total, concurrently with gemcitabine. The initial dose of gemcitabine is 25mg/m² once a week for 6 times. The patients are divided into 9 groups (25mg/m², 50mg/m², 100mg/m², 200mg/m², 300mg/m², 350mg/m², 400mg/m², 450mg/m², 500mg/m²) with 6 patients in each group. Considering about 20% of the cases of dropout, withdrawal, and loss to follow-up in clinical trials, a total of 65 cases are needed in this study. The efficacy is evaluated according to the European Solid Tumor Efficacy Evaluation Standard (RECIST1.1). After induction chemotherapy, radiotherapy, and 3 months after radiotherapy, nasopharyngeal endoscopy and magnetic resonance imaging of the would be reviewed for 1 year, 2 years, and 3 years to evaluate the curative effect. The chest CT, abdominal B-ultrasound, bone scan or PETCT examinations are reviewed to exclud distant metastases. Biopsy diagnosis can be performed for patients suspected of local residual and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing carcinoma (according to WHO histological type)
* Tumor staged as Ⅲ-Ⅳa (according to the 8th AJCC edition staging system)
* Age :18-60
* Performance status: KPS > 70
* Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) < 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) < 2.5×ULN, and bilirubin < ULN
* Renal: creatinine clearance > 60ml/min
* Adequate marrow: leucocyte count > 4×109/L, neutrophil count > 2×109/L, and platelet count > 100×109/L
* Written informed consent

Exclusion Criteria:

* History of allergy to related drugs
* Prior malignancy (except adequately treated carcinoma in-situ of the cervix or basal/squamous cell carcinoma of the skin)
* History of previous RT (except for non-melanomatous skin cancers outside intended RT treatment volume)
* Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerance dose(MTD) | 3 years
  MTD is detemined by the dose that is immediately lower than the dose that produced dose limiting toxicity （DLT）. If DLT occurs in more than half of patients at a certain dose level, the test will be terminated. If DLT occurs in 2 cases,another 6 patients will be treated with this dose. If DLT does not occur in 6 cases, the dose will continue to increase. If it still occurs, the next dose is MTD.

SECONDARY OUTCOMES:
Dose limiting toxicity (DLT) | 3 years
  We determined DLT: a) grade ≥ 3 anemia; b) grade ≥ 3 thrombocytopenia; c) grade ≥ 3 neutropenia no less than 5 days, d) grade 3 febrile neutropenia (absolute neutrophil count < 1.0 x 10^9/L, fever ≥ 38.5℃) despite therapy with granulocyte colony-stimulating factor; and e) any other grades 3-4 toxicity (except alopecia and nausea).
Tumor response rates | 3 years
  Tumor response rate was evaluated according to the RECIST1.1. After induction chemotherapy, radiotherapy and 3 months, 1 year, 2 years, and 3 years of radiotherapy, nasal endoscope and magnetic resonance imaging results were used to evaluate the efficacy. And chest CT scanning, abdominal ultrasound, bone scan or PETCT examination were used to exclude the distant metastases. Pathologic biopsy can be performed for patients who are suspected of locally residual or recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: siyang wang, Principal Investigator — Fifth Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jia WH, Huang QH, Liao J, Ye W, Shugart YY, Liu Q, Chen LZ, Li YH, Lin X, Wen FL, Adami HO, Zeng Y, Zeng YX. Trends in incidence and mortality of nasopharyngeal carcinoma over a 20-25 year period (1978/1983-2002) in Sihui and Cangwu counties in southern China. BMC Cancer. 2006 Jul 6;6:178. doi: 10.1186/1471-2407-6-178. PMID 16822324
- [Background] Zeng Q, Wang J, Lv X, Li J, Yin LJ, Xiang YQ, Guo X. Induction Chemotherapy Followed by Radiotherapy versus Concurrent Chemoradiotherapy in elderly patients with nasopharyngeal carcinoma: finding from a propensity-matched analysis. BMC Cancer. 2016 Aug 30;16(1):693. doi: 10.1186/s12885-016-2661-y. PMID 27577729
- [Background] Meng R, Wei K, Xia L, Xu Y, Chen W, Zheng R, Lin L. Cancer incidence and mortality in Guangdong province, 2012. Chin J Cancer Res. 2016 Jun;28(3):311-20. doi: 10.21147/j.issn.1000-9604.2016.03.05. PMID 27478316
- [Background] Peng G, Wang T, Yang KY, Zhang S, Zhang T, Li Q, Han J, Wu G. A prospective, randomized study comparing outcomes and toxicities of intensity-modulated radiotherapy vs. conventional two-dimensional radiotherapy for the treatment of nasopharyngeal carcinoma. Radiother Oncol. 2012 Sep;104(3):286-93. doi: 10.1016/j.radonc.2012.08.013. Epub 2012 Sep 17. PMID 22995588
- [Background] Zhang MX, Li J, Shen GP, Zou X, Xu JJ, Jiang R, You R, Hua YJ, Sun Y, Ma J, Hong MH, Chen MY. Intensity-modulated radiotherapy prolongs the survival of patients with nasopharyngeal carcinoma compared with conventional two-dimensional radiotherapy: A 10-year experience with a large cohort and long follow-up. Eur J Cancer. 2015 Nov;51(17):2587-95. doi: 10.1016/j.ejca.2015.08.006. Epub 2015 Aug 26. PMID 26318726
- [Background] Huang PY, Zeng Q, Cao KJ, Guo X, Guo L, Mo HY, Wu PH, Qian CN, Mai HQ, Hong MH. Ten-year outcomes of a randomised trial for locoregionally advanced nasopharyngeal carcinoma: A single-institution experience from an endemic area. Eur J Cancer. 2015 Sep;51(13):1760-70. doi: 10.1016/j.ejca.2015.05.025. Epub 2015 Jun 17. PMID 26093812
- [Background] Sun Y, Li WF, Chen NY, Zhang N, Hu GQ, Xie FY, Sun Y, Chen XZ, Li JG, Zhu XD, Hu CS, Xu XY, Chen YY, Hu WH, Guo L, Mo HY, Chen L, Mao YP, Sun R, Ai P, Liang SB, Long GX, Zheng BM, Feng XL, Gong XC, Li L, Shen CY, Xu JY, Guo Y, Chen YM, Zhang F, Lin L, Tang LL, Liu MZ, Ma J. Induction chemotherapy plus concurrent chemoradiotherapy versus concurrent chemoradiotherapy alone in locoregionally advanced nasopharyngeal carcinoma: a phase 3, multicentre, randomised controlled trial. Lancet Oncol. 2016 Nov;17(11):1509-1520. doi: 10.1016/S1470-2045(16)30410-7. Epub 2016 Sep 27. PMID 27686945
- [Background] Chua MLK, Wee JTS, Hui EP, Chan ATC. Nasopharyngeal carcinoma. Lancet. 2016 Mar 5;387(10022):1012-1024. doi: 10.1016/S0140-6736(15)00055-0. Epub 2015 Aug 28. PMID 26321262
- [Background] Ke LR, Xia WX, Qiu WZ, Huang XJ, Yang J, Yu YH, Liang H, Liu GY, Ye YF, Xiang YQ, Guo X, Lv X. Safety and efficacy of lobaplatin combined with 5-fluorouracil as first-line induction chemotherapy followed by lobaplatin-radiotherapy in locally advanced nasopharyngeal carcinoma: preliminary results of a prospective phase II trial. BMC Cancer. 2017 Feb 15;17(1):134. doi: 10.1186/s12885-017-3080-4. PMID 28202000
- [Background] Tang LQ, Chen DP, Guo L, Mo HY, Huang Y, Guo SS, Qi B, Tang QN, Wang P, Li XY, Li JB, Liu Q, Gao YH, Xie FY, Liu LT, Li Y, Liu SL, Xie HJ, Liang YJ, Sun XS, Yan JJ, Wu YS, Luo DH, Huang PY, Xiang YQ, Sun R, Chen MY, Lv X, Wang L, Xia WX, Zhao C, Cao KJ, Qian CN, Guo X, Hong MH, Nie ZQ, Chen QY, Mai HQ. Concurrent chemoradiotherapy with nedaplatin versus cisplatin in stage II-IVB nasopharyngeal carcinoma: an open-label, non-inferiority, randomised phase 3 trial. Lancet Oncol. 2018 Apr;19(4):461-473. doi: 10.1016/S1470-2045(18)30104-9. Epub 2018 Feb 28. PMID 29501366
- [Background] Vanderveken OM, Szturz P, Specenier P, Merlano MC, Benasso M, Van Gestel D, Wouters K, Van Laer C, Van den Weyngaert D, Peeters M, Vermorken J. Gemcitabine-Based Chemoradiation in the Treatment of Locally Advanced Head and Neck Cancer: Systematic Review of Literature and Meta-Analysis. Oncologist. 2016 Jan;21(1):59-71. doi: 10.1634/theoncologist.2015-0246. Epub 2015 Dec 28. PMID 26712958
- [Background] Zhang L, Huang Y, Hong S, Yang Y, Yu G, Jia J, Peng P, Wu X, Lin Q, Xi X, Peng J, Xu M, Chen D, Lu X, Wang R, Cao X, Chen X, Lin Z, Xiong J, Lin Q, Xie C, Li Z, Pan J, Li J, Wu S, Lian Y, Yang Q, Zhao C. Gemcitabine plus cisplatin versus fluorouracil plus cisplatin in recurrent or metastatic nasopharyngeal carcinoma: a multicentre, randomised, open-label, phase 3 trial. Lancet. 2016 Oct 15;388(10054):1883-1892. doi: 10.1016/S0140-6736(16)31388-5. Epub 2016 Aug 23. PMID 27567279
- [Background] Mason KA, Milas L, Hunter NR, Elshaikh M, Buchmiller L, Kishi K, Hittelman K, Ang KK. Maximizing therapeutic gain with gemcitabine and fractionated radiation. Int J Radiat Oncol Biol Phys. 1999 Jul 15;44(5):1125-35. doi: 10.1016/s0360-3016(99)00134-0. PMID 10421547
- [Background] Milas L, Fujii T, Hunter N, Elshaikh M, Mason K, Plunkett W, Ang KK, Hittelman W. Enhancement of tumor radioresponse in vivo by gemcitabine. Cancer Res. 1999 Jan 1;59(1):107-14. PMID 9892194
- [Background] El Deen DA, Toson EA, El Morsy SM. Gemcitabine-based induction chemotherapy and concurrent with radiation in advanced head and neck cancer. Med Oncol. 2012 Dec;29(5):3367-73. doi: 10.1007/s12032-012-0269-x. Epub 2012 Jun 8. PMID 22678924
- [Background] Aguilar-Ponce JL, Granados-Garcia M, Cruz Lopez JC, Maldonado-Magos F, Alvarez-Avitia MA, Arrieta O, Gonzalez-Ramirez I, Lara-Cruz G, Martinez-Juarez I, Medina-Santillan R, Castillo-Hernandez C, De la Garza-Salazar J. Alternating chemotherapy: gemcitabine and cisplatin with concurrent radiotherapy for treatment of advanced head and neck cancer. Oral Oncol. 2013 Mar;49(3):249-54. doi: 10.1016/j.oraloncology.2012.09.008. Epub 2012 Oct 6. PMID 23043985